CLINICAL TRIAL: NCT06975696
Title: Fusion Imaging in Endovascular Thrombectomy for Acute Ischemic Stroke
Acronym: FUSE-IT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Örebro Läns Landsting (Other Government); Helsinki University Central Hospital (Other); University of Turku (Other); Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-08348-01
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Stroke Acute
Keywords: Stroke; endovascular thrombectomy; fusion; interventional neuroradiology; procedure; mTICI
MeSH Terms: conditions — Stroke | interventions — Gene Fusion

STUDY DESIGN:
Intervention Model Description: Multinational, multicenter, prospective, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EVT without Fusion (Active Comparator): Standard endovascular treatment
  Interventions: Procedure: Standard EVT without Fusion
- EVT with Fusion (Experimental): Standard endovascular thrombectomy with Fusion
  Interventions: Procedure: Standard endovascular thrombectomy with Fusion

INTERVENTIONS:
Procedure: Standard endovascular thrombectomy with Fusion — Standard endovacular procedure with the addition of Fusion imaging according to the intended use of the ARTIS Icono Biplane.
  Arms: EVT with Fusion
Procedure: Standard EVT without Fusion — Standard endovacular procedure without the use of Fusion imaging on the ARTIS Icono Biplane.
  Arms: EVT without Fusion

SUMMARY:
Endovascular thrombectomy (EVT) is the standard of care for acute ischemic stroke (AIS) caused by a large vessel occlusion.

Successful recanalization is one of the most important factors for a good patient outcome, especially when obtained within 30 minutes from groin puncture, and the procedural success-rate reaches above 90% at treating centers of excellence. There are however a portion of cases where recanalization is not achieved, which in some cases are attributed to difficult arterial anatomy affecting the ability to catheterize the precerebral target vessel.

In the latest angiography platforms, 3D reconstructions of the aortic, cervical and intracranial arteries from the preprocedural CT angiography can be fused with periprocedural 2D digital subtraction angiography and/or fluoroscopy images, so called 2D/3D Fusion imaging. The preparation steps can be done before patient arrival to the angiography suite and the image fusion can be done in less than a minute during patient preparation. Previous observational studies have shown that the use of fusion imaging during EVT procedures may decrease failed target vessel access and increase procedural success rate and first-pass recanalization rate, without prolonging the procedure.

The purpose of this study is to assess the use of fusion imaging in EVT procedures and its effect on target vessel access, recanalization success-rate and procedure times.

DETAILED DESCRIPTION:
Rationale for the study Successful recanalization is one of the most important factors for a good patient outcome, especially when obtained within 30 minutes from groin puncture, and the procedural success-rate reaches above 90% at treating centers of excellence. In a previously published observational study it was shown that systematic use of Fusion increased the success-rate from 82 to 100%, the first-pass recanalization rate from 49 to 72%, as well as reduced the procedure times.

Risks of study participation The use of Fusion does not require any additional procedure or radiation exposure. A potential risk is that the use of Fusion would prolong the procedure by adding Fusion at the start of the procedure, however in a recently published observational study it was shown that systematic use of Fusion instead reduced the procedure times.

Steps that have be taken to control or mitigate risks. To mitigate the risk that the use of Fusion will cause procedural delays all operators will be trained in using Fusion.

Benefit/risk ratio The use of Fusion has been associated with an increased success-rate from, an increased first-pass recanalization rate and reduced the procedure times. There are no known risks associated with the use of Fusion; therefore, the benefit/risk-ratio is favorable.

Study design This is a multinational, multicenter, prospective, randomized clinical trial.

Study population size The size of the study population is estimated to 300 patients based on a statistical power-estimation (bellow) and the inclusion rate is monitored by the study team on a monthly basis to project the closing of the study.

Data sources Data may be collected from national EVT quality registries, local quality registries, or reported to the study database (RedCAP), depending on local conditions at the including hospital.

Measures to be taken to minimize bias and conflict of interest Monitoring is done by an independent study monitor. Conflicts of interest are reported and disclosed in the publication following the results of the study.

Description of the clinical procedures Fusion on ARTIS icono biplane

In the Icono a previously acquired CT volume (in this study with the preoperative CTA or any previous CTA of the head and neck) can be overlayed (fused) with the live fluoroscopy and digital subtraction angiography (DSA) through the following work-flow:

1. The CTA images are transferred to, or imported from, the Icono.
2. The CTA is opened in the 3D sharing area on the console in the control room.
3. The skeleton is removed using the automated bone removal function.
4. Target structures, such as important vascular landmarks/target vessels can be indicated using the polyline-function.
5. Patients that are awake during the procedure are fixated using a dedicated head holder or by similar measures to minimize head motion after Fusion.
6. At the beginning of the procedure the processed CTA volume is fused using 2D/3D fusion in the Icono.
7. The use of Fusion (or not) should systematically be noted in the procedural report.

   Simultaneous participation in other studies Simultaneous inclusion in other studies that may affect the EVT procedural steps, procedure times or procedural success-rate are not permitted.

   Data collection Data collection is done from local or national quality registries if available, or by direct entering of data in an eCRF tool (RedCAP).

   Lost to follow up A subject will be considered "lost to follow up" and not included in the analysis if they cannot be found in the EPR.

   Imaging core lab An imaging core lab will be set up/used to adjudicate the primary outcome (final recanalization grade according to the mTICI scale).

   Monitoring plan A monitor will be appointed who is independent of the investigational team. Monitoring should be done following the first weeks after study start at a particular study site.

   Remote monitoring is recommended whenever possible. The local PI is responsible for granting access to all relevant source data to the monitor. Access to all relevant source data can be achieved either by direct access to the relevant source data files, including the EVT reports, or by print-outs of the relevant source data files, depending on local circumstances.

   Risk-based monitoring will be used, meaning that the monitoring frequency and scale is adjusted based on the results at previous monitoring. Following the first monitoring occasion, additional monitoring occasions will be initiated by the monitor.

   Statistical design and analysis The statistical design has been done in collaboration with professional statistician at Clinical Trials Sweden - Forum Söder (Dr Sara Jesperson) including statistical power calculation.

   SPSS or R will be used for all statistical analyses. Baseline data will be presented as medians or simple proportions.

   Descriptive statistics will be done for baseline data, safety data and secondary outcome when applicable.

   Primary outcome will be analyzed using 90% confidence interval. Differences between baseline and treatment variables will be explored using chi-squared T-test or Man-Whitney's test. A p-value of <0.05 is considered statistically significant.

   Statistical considerations for sample size In a previous observational study on fusion imaging in EVT, 100% of procedures where fusion imaging was used obtained successful recanalization compared to 86% of procedures performed without fusion imaging.

   When fusion imaging is used within the study, it is reasonable to assume that the recanalization rate may be lower while it may remain similar in the group where fusion imaging is not used.

   Therefore, this study is designed to be able to show a difference in recanalization-rate of 10%, corresponding to 96% success in cases where fusion imaging is used compared to 86% in cases where fusion imaging is not used. With a significance level of 0,05 and 80% power, 128 patients are needed in each group and 256 patients in total. With an expected drop-out frequency of 10%, the study population should be 282 patients.

   Data management The handling of data, including data quality assurance, will comply with regulatory guidelines, including GCP and ISO 14155:2020 and the sponsor's work instructions. All steps and actions taken regarding data management and quality assurance will be according to relevant data handling guidelines.

   A Case Report Form (CRF) can be used to study data. The CRF will be used for data review, data cleaning and issuing and resolving queries. The CRF will be developed and validated using RedCap. The RedCap platform is one of the most used platforms for clinical trials. Each user that will enter data into the CRF will be administered by Lund University, Faculty of Medicine, Library services. Log into the system is done using a secure method of two-factor authentication.

   At the end of the study the CRF data will be merged with data from local- or national quality registries by the professional statistician Sara Jesperson at Clinical Trials Sweden - Forum Söder prior to analysis.

   The CRF data from the subjects will be coded/pseudo-anonymized All adverse event terms recorded on the report forms will be entered into a safety database.

   Personal data is kept to a minimum to minimize the exposure for the study subjects in case of a data breach. Only the date of birth and initials are entered into the eCRF and in the final analysis file, no personal data is included, only coded/pseudonymized data. This minimizes the exposure in case of a data security breach. To minimize the risk of such a breach eCRF data management is done by Lund University.

   Source data will be saved for 10 years as specified in section 3 of chapter III in Annex XV of the MDR on data retention requirements at Skåne University Hospital in Skåne. Region Skåne is responsible for the storage of source data.

   Amendments to the CIP The Investigator should not implement significant changes to the protocol without prior approval by sponsor and prior review and documented approval from the governing Ethics Committee and Competent Authority. The only exception to this requirement is the necessity to eliminate immediate hazards to subjects in the clinical investigation, or when changes involve only administrative aspects (e.g., change in monitors, telephone numbers, etc.).

   In case of changes to the protocol, the investigator will wait for the time specified in article 75 of the MDR or for the approval of the substantial modification, whichever comes first, before implementing the changes.

   Any report of withdrawal of Ethics Committee or Competent Authority approval will be submitted to the Sponsor.

   Deviations from the CIP A protocol deviation is a failure to comply with the requirements of the clinical study as specified in the protocol. Each Investigator shall conduct this clinical study in accordance with the study protocol and any conditions required by the reviewing Ethics Committee and Competent Authority. Deviations from clinical protocol requirements will be reviewed and evaluated on an ongoing basis and, as necessary, appropriate corrective actions put into place.

   The sponsor accepts the right of the Investigator to deviate from the protocol in an emergency when necessary to safeguard the life or the physical well-being of a study subject. The Investigator must give notice of any emergency deviations and justification for the deviation to coordinating center as quickly as possible after the episode, in any event no later than 24-hours after the emergency. The coordinating center will report all deviations to the Ethics Committee and Competent Authority.

   Device accountability Prior to stating the study at a particular site, the sponsor is responsible to ensure that all technical aspects of Fusion are adequate at the participating hospital, as well as relevant training and information has been made available to the operators at the hospital.

   Statements of compliance The clinical investigation will be conducted according to Good Clinical Practice (GCP) guidelines; with informed consent and independent Ethics Committee review and approval as defined in the World Medical Association Declaration of Helsinki, Competent Authority review and approval (if applicable), ISO 14155:2020(E), national legislation, and the Medical Device Regulations (2017/745) of 5 April, 2017.

   This protocol and any amendments will be submitted to a properly constituted Ethics Committee and Competent Authority (if applicable) for formal approval of the study conduct. The decision of the Ethics Committee and Competent Authority (if applicable) concerning the conduct of the study will be made in writing to the Sponsor and a copy of this decision will be provided to the Investigator before commencement of this study.

   The device is CE-marked and the use of the device within the trial are in accordance with the intended use of the CE-mark. All included subjects will be covered by the respective national patient insurance systems.

   Informed consent Informed consent will not be obtained from the included subjects in the study. The rationale for this is that the majority of EVT patients are unable to give written informed consent due to clouded consciousness/clouded mind due to the ongoing stroke, especially those with the most severe stroke. And since this is the most important group to include, the informed consent would introduce a severe selection bias. Informed consent after the procedure would have the same limitation, especially for the patients where the EVT procedure was unsuccessful, and therefore post-EVT informed consent would also introduce a severe selection bias to the study population. Together with the fact that Fusion does not require any additional exposure or procedure to the patients, this is the rationale to not acquire individual informed consent from the participants.

   The Swedish ethical review authority approved the study and waived to need for individual informed consent.

   Adverse event classification and definitions Continuous monitoring of a DSMB/DMC is not done since a previous study indicated very low risk of AEs/SAEs with routine use of Fusion.

   Adverse event (AE) Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs, including an abnormal laboratory finding, in subjects, users or other persons, in the context of a clinical investigation, whether or not related to the investigational device (MDR Article 2(57)).

   Serious Adverse event (SAE)

   A Serious Adverse Event (SAE), as per the European Standard ISO 14155:2020(E), is an AE that led to any of the following:
   1. Death
   2. Serious deterioration in the health of subject, users or other persons as defined by one or more of the following:

      1. a life-threatening illness or injury, or
      2. a permanent impairment of a body structure or body function including chronic diseases, or
      3. in-patient or prolonged hospitalization, or
      4. medical or surgical intervention to prevent life-threatening illness of injury, or permanent impairment to a body structure or body function,
   3. Fetal distress, fetal death, a congenital abnormality or birth defect including physical or mental impairment.

   Planned hospitalization for a pre-existing condition, or a procedure required by the protocol, without serious deterioration in health, is not considered a serious adverse event.

   Adverse device effect (ADE) Any adverse event related to the use of Fusion. AE reporting Any adverse event that occurs during the course of the study must be recorded and reported using the Adverse Event form in the ISF and also recorded in the subject's medical records. These will include events occurring from the point of consent until a subject exits the study. The Investigator must sign each AE report. Investigators must obtain all information available to determine the causality and outcome of the AE and to assess whether it meets the criteria for classification as serious and the relationship of each adverse event to the procedure or device. This determines whether it requires notification to the Sponsor, regulatory agency, and as applicable, EC, within the specified reporting timeframe.

   Pre-existing medical conditions or symptoms occurring prior to the start of the procedure should not be reported as adverse events. In the situation where there is a worsening of a pre-existing medical condition or symptom due to a study related procedure, an adverse event should be reported.

   In the case of any AE, the Investigator shall submit to Sponsor a report within 10 working days after the Investigator first learns of the event.

   The Investigator is required to report all SAEs within 24-hours after first learning of the event to the Sponsor. The primary method of reporting SAEs will be through telephone. Depending upon the nature and seriousness of the adverse event, the Sponsor may request the Investigator to provide anonymous copies of the subject's available supporting documentation (such as the subject's laboratory tests, hospital records, discharge reports, autopsy reports, Investigator summaries, etc.) to document the adverse event. The Sponsor is responsible in Europe for ensuring that the required and adequate information concerning the reported SAE is relayed to the appropriate Competent Authority using the MEDDEV 2.7/3 SAE Report Table. All other adverse events (i.e., other than serious adverse events) must be recorded on the appropriate adverse event eCRF.

   Sponsor, in cooperation with the Investigator, will assess all serious adverse events for potentially reporting to the Regulatory Authorities and EC.

   For any adverse event that is ongoing at the time of the initial report, periodic follow-up information is required until the adverse event is resolved or is judged to be chronically stable, or until the conclusion of the study for the subject. The site should submit relevant follow-up information related to the adverse event as soon as it is available.

   Contact details for reporting serious adverse events and serious adverse device effects Dr Johan Wasselius Department of Radiology, Interventional Neuroradiology Department of Clinical Sciences Lund, Lund University Phone: ‭+46 70173994‬3, +46 46173083 E-mail: johan.wasselius@skane.se End, suspension, or premature termination of the study The study ends 3 months after inclusion of the last included patient. The principal investigator, EC, or regulatory authority may suspend or prematurely terminate participation in the clinical research at the Investigation sites for which they are responsible.

   Any signs of unknown or increased risks for the subjects will be discussed by the sponsor and investigator to assess the impact on the subjects and clinical research. If suspicion of an unacceptable risk to subjects arises during the clinical research, or when so instructed by the EC or regulatory authorities, the sponsor shall suspend the clinical research while the risk is assessed.

   The sponsor shall terminate the clinical research if an unacceptable risk is confirmed.

   If suspension or premature termination occurs, the terminating party shall justify its decision in writing and promptly inform the other parties with whom they are in direct communication. The principal investigator and sponsor shall keep each other informed of any communication received from either the EC or the regulatory authority.

   Serious or repetitive occurrence of deviations from study protocol or non-compliance with regulations may also be reason for early termination or suspension of a study site.

   Publication policy The clinical investigation will be registered in a publicly available database (Clintrials.gov).

   The results of the clinical investigation will be made publicly available. The results of the clinical investigation will be offered for publication within one year of the end of the study. The PI is responsible for this work. All investigators that contributed to the content of the publication should be included in the author list.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Eligible for an EVT procedure

Exclusion Criteria:

1. Previous inclusion in this study
2. No access to a preoperative CTA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful recanalization | At the end of the EVT procedure
  Defined as modified Treatment in Cerebral Infarction score (mTICI) 2b or better.

SECONDARY OUTCOMES:
Target vessel access | During the EVT procedure
  Successful catheterization of the precerebral target vessel
Excellent recanalization | At the end of the procedure
  Final recanlization grade defined as mTICI 2c or better
First pass recanalization | At the end of the procedure
  Successful recanalization on the first thrombectomy attempt.
Time from groin puncture to precerebral target vessel access | During the procedure
  Defined as the time of the first angiography from the precerebral target vessel.
Time from groin puncture to first pass with stent-retriever and/or direct aspiration. | During the procedure.
  Defined at time from groin puncture to the first deployment of a stent-retriever or the first direct aspiration.
Time from groin puncture to recanalization | During the procedure.
  Defined as the time from groin puncture to recanalization grade 2B or better is obtained. If successful recanalization is not obtained during the procedure, the time of the final angiogram is used.
Groin to first-pass recanalization within within 30 minutes | During the procedure.
  Defined as whether first-pass recanalization within 30 minutes of groin-time is obtained or not.
Successful image fusion | During the procedure.
  Defined as whether successful Fusion is performed during the procedure or not.

OTHER OUTCOMES:
Perioperative death | During the procedure.
  If the patient dies during the procedure or not.
Vessel perforation | During the procedure.
  Any intracranial vessel perforation with observed contrast extravasation on DSA.
Vessel dissection | During the procedure.
  Any iatrogenic arterial dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Andersson, MSc, Study Director — Lund University; Johan Wasselius, MD, PhD, Principal Investigator — Skåne University Hospital and Lund University
Locations (3):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Turku University Hospital, Turku
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
Personal data of the participants may not be shared. An aggregated dataset supporting the conclusions of the study may be shared upon resonable request including necessary permits.

REFERENCES:
- [Result] Fusion Imaging in Endovascular Thrombectomy for Acute Ischemic Stroke. Lovisa Landström, Emma Hall, Björn Hansen and Johan Wassélius. Stroke: Vascular and Interventional Neurology. Online ahead of print. doi: 10.1161/SVIN.124.001636
- [Result] Ribo M, Flores A, Rubiera M, Pagola J, Mendonca N, Rodriguez-Luna D, Pineiro S, Meler P, Alvarez-Sabin J, Molina CA. Difficult catheter access to the occluded vessel during endovascular treatment of acute ischemic stroke is associated with worse clinical outcome. J Neurointerv Surg. 2013 May;5 Suppl 1:i70-3. doi: 10.1136/neurintsurg-2012-010438. Epub 2012 Oct 31. PMID 23117130
- [Result] Snelling BM, Sur S, Shah SS, Chen S, Menaker SA, McCarthy DJ, Yavagal DR, Peterson EC, Starke RM. Unfavorable Vascular Anatomy Is Associated with Increased Revascularization Time and Worse Outcome in Anterior Circulation Thrombectomy. World Neurosurg. 2018 Dec;120:e976-e983. doi: 10.1016/j.wneu.2018.08.207. Epub 2018 Sep 6. PMID 30196176
- [Result] Penide J, Mirza M, McCarthy R, Fiehler J, Mordasini P, Delassus P, Morris L, Gilvarry M. Systematic Review on Endovascular Access to Intracranial Arteries for Mechanical Thrombectomy in Acute Ischemic Stroke. Clin Neuroradiol. 2022 Mar;32(1):5-12. doi: 10.1007/s00062-021-01100-7. Epub 2021 Oct 12. PMID 34642788
- [Result] Lajthia O, Almallouhi E, Ali H, Essibayi MA, Bass E, Neyens R, Anadani M, Chalhoub R, Kicielinski K, Lena J, Porto G, Sattur M, Spiotta AM, Kasab SA. Failed mechanical thrombectomy: prevalence, etiology, and predictors. J Neurosurg. 2023 Jan 20;139(3):714-720. doi: 10.3171/2022.12.JNS222152. Print 2023 Sep 1. PMID 36670537
- [Result] Wasselius J, Hall E, Ramgren B, Andersson T, Ullberg T. Procedural factors associated with successful recanalization in patients with acute ischemic stroke treated with endovascular thrombectomy-a nationwide register-based observational study. Interv Neuroradiol. 2024 Apr 22:15910199241248268. doi: 10.1177/15910199241248268. Online ahead of print. PMID 38646674
- [Result] Fischer U, Kaesmacher J, Strbian D, Eker O, Cognard C, Plattner PS, Butikofer L, Mordasini P, Deppeler S, Pereira VM, Albucher JF, Darcourt J, Bourcier R, Benoit G, Papagiannaki C, Ozkul-Wermester O, Sibolt G, Tiainen M, Gory B, Richard S, Liman J, Ernst MS, Boulanger M, Barbier C, Mechtouff L, Zhang L, Marnat G, Sibon I, Nikoubashman O, Reich A, Consoli A, Lapergue B, Ribo M, Tomasello A, Saleme S, Macian F, Moulin S, Pagano P, Saliou G, Carrera E, Janot K, Hernandez-Perez M, Pop R, Schiava LD, Luft AR, Piotin M, Gentric JC, Pikula A, Pfeilschifter W, Arnold M, Siddiqui AH, Froehler MT, Furlan AJ, Chapot R, Wiesmann M, Machi P, Diener HC, Kulcsar Z, Bonati LH, Bassetti CL, Mazighi M, Liebeskind DS, Saver JL, Gralla J; SWIFT DIRECT Collaborators. Thrombectomy alone versus intravenous alteplase plus thrombectomy in patients with stroke: an open-label, blinded-outcome, randomised non-inferiority trial. Lancet. 2022 Jul 9;400(10346):104-115. doi: 10.1016/S0140-6736(22)00537-2. PMID 35810756
- [Result] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Result] Jang KM, Choi HH, Nam TK, Byun JS. Clinical outcomes of first-pass effect after mechanical thrombectomy for acute ischemic stroke: A systematic review and meta-analysis. Clin Neurol Neurosurg. 2021 Dec;211:107030. doi: 10.1016/j.clineuro.2021.107030. Epub 2021 Nov 11. PMID 34823155
- [Result] Alawieh A, Pierce AK, Vargas J, Turk AS, Turner RD, Chaudry MI, Spiotta AM. The golden 35 min of stroke intervention with ADAPT: effect of thrombectomy procedural time in acute ischemic stroke on outcome. J Neurointerv Surg. 2018 Mar;10(3):213-220. doi: 10.1136/neurintsurg-2017-013040. Epub 2017 May 2. PMID 28465405